CLINICAL TRIAL: NCT03135990
Title: Using Virtual Reality in Exposure-Based Treatment for Social Anxiety in Youth
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to the start of the COVID-19 pandemic.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1701017878
Record Dates: First submitted 2017-03-21; First posted 2017-05-02 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Social Anxiety; Social Anxiety Disorder; Social Anxiety Disorder of Childhood
Keywords: Virtual Reality; Exposure Therapy; Cognitive Behavioral Therapy; Extinction Learning
MeSH Terms: conditions — Phobia, Social | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Cognitive Behavioral Therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT + VR (Experimental): Cognitive Behavioral Therapy with Virtual Reality technology.
  Interventions: Behavioral: Cognitive Behavioral Therapy with Virtual Reality Technology

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy with Virtual Reality Technology — Cognitive Behavioral Therapy Intervention: This manualized intervention is a modified version of the Unified Protocol for Emotional Disorders in Youth, a modular Cognitive Behavioral Therapy protocol for anxiety disorders and depression with demonstrated efficacy in youth. The 10-session intervention includes psychoeducation about anxiety disorders and their treatment (1 session), emotion awareness and regulation (2 sessions), exposure therapy using virtual reality environments (6 sessions), and review and relapse prevention (1 session). All treatment sessions will be videotaped to ensure fidelity to treatment manual and modules.

SUMMARY:
Anxiety disorders are the most common mental health diagnosis in the US and are associated with avoidance that causes functional impairments and decreases quality of life. Social anxiety disorder is among the most prevalent anxiety disorders, with most common age of onset being in adolescence. The frontline treatment for social anxiety disorder is cognitive behavioral therapy with exposure. However, a significant number of adolescent patients do not get better after completing cognitive behavioral therapy or experience relapse. This could be explained by findings in both mice and humans suggesting that cue-based extinction learning occurs less readily in adolescents than in children and adults. Studies using mouse-models have overcome this age disparity by enhancing contextual cues when fear extinction learning takes place. Providing realistic learning contexts for exposure could be the key to enhancing treatment effects in adolescents. This is often challenging for a variety of reasons, including difficulty realistically mimicking anxiety-provoking social situations due to limited resources, clinician training, time, or motivation. Virtual reality environments could provide contextual exposures for social anxiety.

This pilot study will test the feasibility of integrating virtual reality technology in exposure-based treatment in youth ages 13-23 diagnosed with social anxiety disorder with the goal of approximating equivalent efficacy with traditional cognitive behavioral therapy, and assessing feasibility of virtual reality technology with this population. We will also pilot a fear conditioning and extinction learning paradigm to explore the relationship between extinction learning and efficacy of virtual reality exposure therapy, using physiological assessment indicators to mark changes in fear response. These markers will also be used prior to the initiation of the therapy to assess the degree to which virtual reality environments invoke a true fear response, comparing the 12 participants with social phobia to 12 age matched, non-anxious control participants. The aims of this study are threefold: to assess feasibility of using virtual reality in treatment of social anxiety in youth, to examine whether virtual reality invokes arousal similar to anxiety and test the physiological assessment protocol, and to evaluate whether exposure using virtual reality environments reduces symptoms of social anxiety and related functional impairment.

DETAILED DESCRIPTION:
Lifetime prevalence of social anxiety disorder in adolescents is estimated to be 8.6%, with the most common age of onset being ages 15-17. Social anxiety disorder is related to significant functional impairment and, if untreated, puts youth at risk for depression and substance abuse, and results in failure to meet important academic, social, and occupational milestones. The current literature supports cognitive behavioral therapy with exposure therapy, selective serotonin re-uptake inhibitor medications, and their combination for the treatment of anxiety disorders with good effects. However, even with gold standard treatment, a significant number of patients do not get better or experience relapse. Exposure therapy is based on the principles of fear extinction, such that cues associated with threat are presented in a safe and controlled way until they are experienced as safe and fear responses are reduced. Studies in mice and non-anxious humans have demonstrated cue-based fear extinction learning to be less robust in adolescence than it is in childhood or adulthood. However, mouse-models suggest that context-based extinction learning closes the gap between age-groups, with adolescents performing as well on extinction learning tasks when put back in the original environment where the fear was acquired.

Similarly, clinical research suggest that exposure therapy is most useful when exposures are conducted in the same or similar environments to where the fear is experienced in everyday life. However, there are many barriers to providing contextual based exposure therapy, particularly for social anxiety, including paucity of well-trained exposure therapists in many areas of the country, and difficulty generating or accessing realistic social situations for convincing exposures.

Virtual reality offers a promising avenue for contextual exposures, by increasing the availability of certain contexts that cannot be readily mimicked in therapy. Furthermore, in vivo exposure situations can feel overwhelming for some individuals (patients and therapists), resulting in refusal to engage in exposure altogether. Virtual reality technology could allow for more gradual titration of exposure for those patients that require lower intensity exposures, and can be done in the therapy office for clinicians who do not have the time, resources, experience, or comfort level to travel outside of their office in pursuit of appropriate exposure environments. Even for seasoned exposure therapists, virtual reality could serve as a practice step in preparation for in vivo exposures or could be used in lieu of in vivo exposures if necessary. There has been extensive research on the use of virtual reality in facilitating exposure in a variety of populations. However, its effectiveness has not been demonstrated in adolescents with social phobia, and research is limited in adolescent samples in general.

The pilot study proposed for this National Alliance for Research on Schizophrenia and Depression award would test the overall hypothesis that virtual reality technology is feasible, acceptable, and will enhance exposure-based therapy for socially anxious youth. Studies will be focused on testing the feasibility of integrating virtual reality technology into exposure-based treatment in adolescents and young adults (ages 13-23) diagnosed with social anxiety disorder with the goal of approximating equivalent efficacy with traditional cognitive behavioral therapy, and assessing feasibility, usability, and acceptability of the virtual reality technology with this population. In addition, we would pilot a fear conditioning and extinction learning paradigm with the subjects to explore the relationship between extinction learning and efficacy of virtual reality exposure therapy, using physiological assessment indicators to mark changes in fear response, including skin conductance, heart rate, heart rate variability, and startle. These physiological markers would also be used prior to the initiation of the therapy to assess the degree to which the virtual reality environments invoke a true fear response, comparing the 12 subjects with social phobia to 12 age-matched, non-anxious control subjects. If feasible and effective, these procedures would be used for a larger future study, and pilot data would be used for a K-award, R21, or R01 grant application, including neuroimaging to learn more about the neural circuitry involved in fear learning via virtual reality technology.

SPECIFIC AIMS

Specific Aim 1: To assess the feasibility, acceptability, and usability of simulated exposure using virtual reality environments in treatment of social anxiety in youth ages 13-23.

Hypothesis: We hypothesize that the use of this technology will be feasible, evidenced by 75% completion of the treatment protocol.

Specific Aim 2: To examine the degree to which virtual reality environments invoke arousal consistent with anxiety, and test the feasibility, acceptability, and usability of psychophysiological assessment protocol.

Hypothesis: We hypothesize that subjects will exhibit elevated arousal during virtual reality-assisted exposures, evidenced by increased skin conductance, heart rate, and startle response, and expect the procedures to be feasible and acceptable as evidenced by high completion and low drop out.

Specific Aim 3: To evaluate the impact of simulated exposure using virtual reality environments in reducing symptoms of social anxiety and related functional impairment.

Hypothesis: We hypothesize that subjects will exhibit a decrease in anxiety evidenced by reduction in Anxiety Disorders Interview Schedule Clinician Severity Rating ≤ 4 and improvement in global functioning evidenced by Clinical Global Impression- Improvement rating ≤ 3.

METHODS

Study Design: 12 adolescents and young adults (ages 13- 23) with social anxiety disorder (cognitive behavioral therapy + virtual reality), and 12 age-matched comparison subjects (Controls) will be recruited for participation in this pilot feasibility study. Subjects on psychiatric medication must be on a stable dose for at least 2 months prior to study participation and remain symptomatic to the level identified for inclusion in the cognitive behavioral therapy + virtual reality group (Anxiety Disorders Interview Schedule Clinician Severity Rating ≥ 4). Controls must not meet criteria for any anxiety disorder. Control subjects will not complete the intervention, but will participate solely in the initial virtual reality arousal test and the fear extinction paradigm.

Assessment measures: Clinician administered measures include the Anxiety Disorder Interview Schedule for DSM 5 to determine initial diagnostic status. The Clinical Global Impression Scale (CGI) will assess overall symptom severity and improvement. Self-report measures include the Screen for Child Anxiety Related Disorders and the World Health Organization Disability Scale-12 assessment of global functioning. Subjects in the virtual reality + cognitive behavioral therapy group will complete these measures at pre-treatment, at post-treatment, and at 3 month follow up. Controls will complete these measures at only one time point.

Virtual Reality technology: virtual reality simulation allows subjects wearing a head-mounted display to view computer-generated 3-D imagery of a variety of social environments which evoke distress in individuals diagnosed with social anxiety. Subjects report on distress levels throughout the exercise.

Cognitive Behavioral Therapy Intervention: The manualized cognitive behavioral therapy intervention used in this study will be a modified version of the Unified Protocol for Emotional Disorders in Youth (UP-Y), which is a modular cognitive behavioral therapy protocol for anxiety disorders and depression with demonstrated efficacy in youth. The modular approach allows for patient engagement in exposure therapy at earliest readiness, and also allows for the structured implementation of other cognitive behavioral therapy components. The 10-session intervention includes psychoeducation about anxiety disorders and their treatment (1 session), emotion awareness and regulation (2 sessions), exposure therapy using virtual reality environments (6 sessions), and review and relapse prevention (1 session). All treatment sessions will be videotaped to ensure fidelity to treatment manual and modules.

Psychophysiological measures: The Biopac system will measure physiological arousal through measures of skin conductance, heart rate, heart rate variability, and startle response (via eye blink reflex). Each of the tests involved in collection of biological measures is a standard, non-painful and non-invasive procedure.

Fear Conditioning & Extinction Paradigm: Subjects will participate in a laboratory test of extinction training during their initial assessment in order to establish extinction learning as a potential predictive marker of treatment outcome. Subjects will be exposed to two shapes on a computer screen, one shape (conditioned stimulus; CS+) will be paired with an aversive stimulus (unconditioned stimulus) on 38% of the trials, whereas the other shape will never be paired with aversive stimulus (conditioned stimulus-). Later, they will undergo extinction training in which the two conditioned stimuli will be repeatedly presented without the unconditioned stimulus. Extinction will be measured as the difference score of skin conductance response to the conditioned stimulus+ and conditioned stimulus-.

ELIGIBILITY:
Inclusion Criteria for Virtual Reality/CBT Group:

1. Ages 13-23 with a primary diagnosis of social anxiety disorder.
2. Anxiety Disorders Interview Schedule-5 Clinician Severity Rating greater than 4
3. IQ estimate of 70 or higher.
4. Comorbid disorder (e.g., Attention Deficit Hyperactivity Disorder, Obsessive Compulsive Disorder, Oppositional Defiant Disorder) will be allowed provided that the anxiety symptoms are of primary concern to parents and comorbid symptoms are not of sufficient severity to require immediate treatment other than that provided by the current study.
5. Sufficient command of the English language to comply with study protocol.
6. Participants on psychiatric medication must be on a stable dose for at least 2 months prior to study participation and remain symptomatic to the level identified for study inclusion (Anxiety Disorders Interview Schedule-5 less than or equal to 4). Family agrees to refrain from med changes over the course of the study if at all possible.

Inclusion Criteria for Control Group:

1. Ages 13-23.
2. Does not meet criteria for anxiety or mood disorder on Anxiety Disorders Interview Schedule-5.

Exclusion Criteria:

1. Unable to consent.
2. A prior or present diagnosis of receptive and expressive language disorder and/or pervasive developmental disorder or severe mental retardation.
3. Current substance use disorder or dependence as primary diagnosis.
4. Recent suicide behavior (last month) or any other psychiatric condition that requires more intensive care (e.g., psychotic episode, manic episode).
5. Youth or parent/third party not fluent in English.

Ages: 13 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Change in diagnostic in diagnostic status and severity of social anxiety symptoms measured by ADIS | Initial Visit,Immediately after the intervention, and Three Month Follow Up Visit
  Anxiety Disorders Interview Schedule is used to assess change in diagnostic status and severity of social anxiety symptoms. A low score of a 3 or below would be a sub-clinical representation of the disorder, a 4 represent moderate severity and a high score of 5-8 would be a clinically severe representation of the disorder.

SECONDARY OUTCOMES:
Change in depression and suicidality as measured by CESD-R | Initial Visit, Immediately after the intervention, and Three Month Follow Up Visit
  Center for Epidemiologic Studies Depression Scale will be used to measure change of depression and suicidality. Based on how CESD-R is answered, patients are determined to meet criteria for one of 5 categories: Major Depressive Episode; Probable Major Depressive Episode; Possible Major Depressive Episode; Subthreshold depression symptoms; No clinical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Pelcovitz, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No